CLINICAL TRIAL: NCT04330651
Title: Outcomes' Predictors in Post-Surgery Extracorporeal Life Support
Brief Title: Post-Surgery Extracorporeal Life Support
Acronym: PC-ECLS
Status: Recruiting | Type: Observational
Sponsor: University of Florence (Other)
Collaborators: Sandro Gelsomino (Unknown); Edvin Prifti (Unknown); Francesco Cabrucci (Unknown); Marco Bugetti (Unknown); Orlando Parise (Unknown); Aleksander Dokollari (Unknown)
Responsible Party: Principal Investigator, Massimo Bonacchi, Professor, University of Florence
Other Study IDs: PC-ECLS Study
Record Dates: First submitted 2020-03-19; First posted 2020-04-01 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Cardiogenic Shock; Extracorporeal Life Support; Extracorporeal Membrane Oxygenation Complication; Post Cardiac Arrest Syndrome; Post-cardiac Surgery
Keywords: extracorporeal life support; ecls; ecmo; outocome; prognostic factors; extracorporeal membrane oxygenation
MeSH Terms: conditions — Shock, Cardiogenic; Post-Cardiac Arrest Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: ECLS — Emergency application of Extracorporeal Life Support in post-surgical patients

SUMMARY:
Extracorporeal Life Support (ECLS) may provide pulmonary and circulatory support for patients with acute heart failure refractory to conventional medical therapy. However, indications and effectiveness of ECLS engagement post-surgery remains a concern. The investigators sought to analyze indications, modality and outcomes of PS-ECLS, to identify predictors of early and midterm survival after PS-ECLS. The investigators have recorded prospectively, and analysed data of 209 consecutive PS-ECLS patients between January 2004 and December 2018. Demographic and clinical data before, during and after PS-ECLS were collected and their influence on hospital mortality and outcomes (early and midterm) will analyse. Multivariate analysis of pre PS-ECLS implantation factors (as age, female sex , insulin-dependent diabetes, pulmonary hypertension, STS, type of surgical procedure data, pre-ECLS blood lactate level) will be made for identify prognostic risk factors of in-hospital mortality. Overall survival will be analysed, at 6 months,1-year and 5-years, respectively and the factors influencing mild/term outcome will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent cardiac surgery

Exclusion Criteria:

* Age < 18 years

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients underwent cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2004-01; Primary Completion 2021-03-19 (Actual); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 1 month after surgery
  Evaluate Early, mid and late Survival
Survival | At 1 Year after surgery
  mid-time survival
Survival | At 5 years after surgery
  late survival

SECONDARY OUTCOMES:
Prognostic factors | Early: 1 month after surgery
  Identify early and late negative and positive prognostic factors
Prognostic Factors | Late: 5 years after surgery
  Identify early and late negative and positive prognostic factors

CONTACTS AND LOCATIONS:
Locations (1):
- Massimo Bonacchi, Florence, Italy